CLINICAL TRIAL: NCT04187235
Title: Laparascopic Keyhole vs Sugarbaker Repair in Parastomal Hernia: A Long Term Case-controlled Prospective Study of Consecutive Patients.
Brief Title: Laparascopic Keyhole vs Sugarbaker Repair in Parastomal Hernia
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Vitaly Alexandrovich Gameza, MD, Aalborg University Hospital
Other Study IDs: Keyhole vs Sugarbaker
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Parastomal Hernia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Keyhole rapair: 74 patients who undervent parastomal hernia repair with keyhole technique 1997-2009
  Interventions: Procedure: Laparascopic repair of parastomal hernia
- Sugarbaker repair: 61 patients who undervent parastomal henia repair a.m. Sugarbaker 2009-2015
  Interventions: Procedure: Laparascopic repair of parastomal hernia

INTERVENTIONS:
Procedure: Laparascopic repair of parastomal hernia — Laparascopic repair of parastomal hernia

SUMMARY:
This is a non-randomised case-controlled prospective study of consecutive patients with parastomal hernia, comparing the laparoscopic Keyhole repair with the modified Sugarbaker repair.

DETAILED DESCRIPTION:
Objective: To compare the laparoscopic Keyhole repair with the modified Sugarbaker repair in a nonrandomised case-controlled prospective study of consecutive patients with parastomal hernia.

Summary Background Data: Two reviews of uncontrolled studies concluded that the Sugarbaker repair is superior to the Keyhole repair. The present study challenges the claim.

Methods: In two time periods 135 patients with a parastomal hernia were repaired with the Keyhole technique (74 patients, using a two-layer mesh of polypropylene and ePTFE with a self-cut slit, 1997- 2009) or the Sugarbaker technique (61 patients, using a coated polypropylene mesh, 2009-2015). The patients in the two groups matched with regard to age, gender, ASA score, colostomy or ileostomy hernia, previous repairs, size of fascial defect and simultaneous repair of a concurrent incisional hernia. Observation time was defined as time to recurrence, stoma re-siting, mesh removal, death, or last non-event visit

ELIGIBILITY:
Inclusion Criteria: Patients with a diagnosis of parastomal hernia and indication for surgical treatment -

Exclusion Criteria: None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with parastomal hernia referred to Aarhus University Hospital
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Recurrence | 3 years
  Recurrence of parastomal hernia

SECONDARY OUTCOMES:
Mesh-related morbidity | 3 years
  Late mesh-related morbidity
Postoperative complications | 30 days after surgery
  Early postoperative complication

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wara, DMSc, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
We have no permission to share individual participant data with 3rd parties